CLINICAL TRIAL: NCT01842113
Title: Quality of Life and Nutritional Improvements in Cirrhotic Patients Following Hepatic Encephalopathy Using Rifaximin.
Brief Title: Quality of Life and Nutritional Improvements in Cirrhotic Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI Initiated study - PI left facility
Sponsor: Tampa General Hospital (Other)
Responsible Party: Principal Investigator, Guy Neff, MD, Medical Doctor, Tampa General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rifaximin and Nutrition
Record Dates: First submitted 2013-04-11; First posted 2013-04-29 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Liver Cirrhosis; Hepatic Encephalopathy; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy; Hypertension, Portal | interventions — Rifaximin; Lactulose; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactulose and Rifaximin Placebo (Active Comparator): Standard portal hypertension care, standard nutritional advice, Lactulose 30ml three times a day and Rifaximin (Xifaxan) Placebo twice a day.
  Interventions: Drug: Lactulose; Drug: Rifaximin Placebo
- Rifaximin and Lactulose Placebo (Active Comparator): Rifaximin (Xifaxan) twice a day and Lactulose Placebo three times a day.
  Interventions: Drug: Rifaximin; Drug: Lactulose Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 550mg by mouth twice a day
  Other Names: Xifaxan
  Arms: Rifaximin and Lactulose Placebo
Drug: Lactulose — Lactulose 30ml by mouth three times a day
  Other Names: Enulose; Generlac; Cholac; Constulose; Kristalose; Laxilose; Portalac; Hepatalac; Constilac
  Arms: Lactulose and Rifaximin Placebo
Drug: Lactulose Placebo — Lactulose Placebo 30ml three times a day
  Arms: Rifaximin and Lactulose Placebo
Drug: Rifaximin Placebo — Rifaximin Placebo twice a day
  Other Names: Sugar Pill
  Arms: Lactulose and Rifaximin Placebo

SUMMARY:
The purpose of this study is to determine whether taking Rifaximin (Xifaxan) in conjunction with the use of nutritional concepts is effective in improving morbidity and quality of life in cirrhotic patients suffering from hepatic encephalopathy (HE).

DETAILED DESCRIPTION:
Prevention of portal hypertension complications should be at the forefront. In doing so, the end result will be an improvement in the multitude of morbidity and mortality issues. The proposed prospective trial will compare patients with similar demographics and medical and clinical settings utilizing standard of care therapy. Study subjects will be randomly assigned into two treatment groups. Group one will receive Lactulose 30ml three times a day as SOC and Rifaximin Placebo 550mg twice a day with nutritional supervision and group two will receive Rifaximin 550mg twice per day as SOC and Lactulose placebo 30ml three times per day with nutritional supervision.

ELIGIBILITY:
Inclusion Criteria:

* Male and female gender of Age 18 years or older
* Liver cirrhosis defined as one or more of the following: Radio-graphically proven portal hypertension (CT with nodular appearance) or Liver biopsy with cirrhosis
* Model for End Stage Liver Disease (MELD) score < 20
* Willingness to provide written informed consent, and participate in all study requirements
* Sodium greater than 130 meq/L
* Conn Score < 2

Exclusion Criteria:

* Active alcohol consumption
* Serum total bilirubin level > 5 mg/dl
* History of hepatocellular carcinoma (HCC) and malignancies other than basal cell carcinoma of the skin
* Pregnant or breastfeeding women
* Subject has renal insufficiency requiring routine dialysis
* Poorly controlled diabetes as defined by HgA1C > 10
* Narcotic/psychotropic usage other than a stable dose of antidepressant and/or methadone. Neurontin (gabapentin) and Lyrica (pregabalin) are permitted if the subject has been on a stable dose for at least 2 months prior to the screening visit and no change of dosing is expected throughout the length of the trial
* Any of the following diagnoses:
* HIV
* Evidence of severe concomitant illness or any condition that makes them unsuitable for the study in the opinion of the investigator(s)
* Subject has received an investigational drug within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Outcomes of Change in Quality of Life Assessment Between the Two Groups | Participants will be followed for 180 days
  Quality of Life will be determined by the Chronic Liver Disease Foundation Questionnaire (CLDQ), the Sleep Scale by Hays, R.D.&Stewart, A.L. and the Multidimensional Assessment of Fatigue (MAF) Scale and measured based upon Subjective Global Assessment (SGA).
Nutritional Improvement Between the Two Groups | Participants will be followed for 180 days
  These outcomes will be determined as Body Composition Analysis via the Quadscan 4000 BIA device manufactured by Bodystat;calories burned, steps taken and levels of physical activity to sleep efficiency will be measured via the Bodymedia CORE Fit actigraph device and various standard of care laboratories.

SECONDARY OUTCOMES:
Markers of improvement in general health | Participants will be followed for 180 days
  These outcomes will be determined as Body Composition Analysis via the Quadscan 4000 BIA device manufactured by Bodystat;calories burned, steps taken and levels of physical activity to sleep efficiency will be measured via the Bodymedia CORE Fit actigraph device and various standard of care laboratories.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Neff, MD, MBA, Principal Investigator — Tampa General Medical Group
Locations (1):
- Tampa General Medical Group, Tampa, Florida, United States